CLINICAL TRIAL: NCT03272295
Title: A Randomised, Controlled, Double-Blind Study to Examine Nicotine Pharmacokinetics and Smoking Behaviour in Healthy Smokers When Smoking Cigarettes Containing Different Commonly Used Ingredients
Brief Title: A Nicotine Pharmacokinetics and Smoking Behaviour Study Examining Cigarette Ingredients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British American Tobacco (Investments) Limited (Industry)
Collaborators: Philip Morris Products S.A. (Industry); Imperial Brands PLC (Industry); Japan Tobacco Inc. (Industry); Korea Ginseng Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: BAT1117009; CA21208 (Other: Celerion GB Ltd)
Record Dates: First submitted 2017-08-15; First posted 2017-09-05 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Healthy Volunteers; Smoking
MeSH Terms: conditions — Smoking | interventions — Tobacco Products; Chocolate; fenugreek seed meal; Glycerol; Guaiacol; Propylene Glycol; Sorbitol

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: A double-blind study in respect of the site (except pharmacy) and subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Reference product (product 1) x 2, Single ingredients products 2, 3, 4, 5, 6 and Multiple ingredient product (product 12). Single cigarette each for nicotine PK assessment and smoking behaviour assessment.
  Interventions: Other: Reference cigarette; Other: Cigarette with carob bean extract; Other: Cigarette with cocoa powder; Other: Cigarette with fenugreek extract; Other: Cigarette with fig juice; Other: Cigarette with glycerol; Other: Cigarette with multiple ingredients
- Arm B (Experimental): Reference product (product 1), Single ingredients products 7, 8, 9, 10, 11 and Multiple ingredient product (product 12). Single cigarette each for nicotine PK assessment and smoking behaviour assessment.
  Interventions: Other: Reference cigarette; Other: Cigarette with guaiacol; Other: Cigarette with liquorice extract powder; Other: Cigarette plus I-menthol; Other: Cigarette with propylene glycol; Other: Cigarette with sorbitol; Other: Cigarette with multiple ingredients

INTERVENTIONS:
Other: Reference cigarette — The reference product is based on a commercially-available king-size cigarette design (length 83 mm, circumference 24.6 mm) with a single segment cellulose acetate filter and tobacco blend recipe without ingredients.
Other: Cigarette with carob bean extract — Based on reference cigarette with added ingredient
  Arms: Arm A
Other: Cigarette with cocoa powder — Based on reference cigarette with added ingredient
  Arms: Arm A
Other: Cigarette with fenugreek extract — Based on reference cigarette with added ingredient
  Arms: Arm A
Other: Cigarette with fig juice — Based on reference cigarette with added ingredient
  Arms: Arm A
Other: Cigarette with glycerol — Based on reference cigarette with added ingredient
  Arms: Arm A
Other: Cigarette with guaiacol — Based on reference cigarette with added ingredient
  Arms: Arm B
Other: Cigarette with liquorice extract powder — Based on reference cigarette with added ingredient
  Arms: Arm B
Other: Cigarette plus I-menthol — Based on reference cigarette with added ingredient
  Arms: Arm B
Other: Cigarette with propylene glycol — Based on reference cigarette with added ingredient
  Arms: Arm B
Other: Cigarette with sorbitol — Based on reference cigarette with added ingredient
  Arms: Arm B
Other: Cigarette with multiple ingredients — Based on reference cigarette plus propylene glycol, glycerol, liquorice extract powder, cocoa powder, carob bean extract, fig juice concentrate, maltol, guaiacol, geraniol, fenugreek extract.

SUMMARY:
This study will compare nicotine delivery and smoking behaviour in healthy subjects using several combustible cigarette prototypes containing different ingredients which are commonly used in the European Union.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be:

   1.1. males or females 1.2. 21 to 55 years of age, inclusive, demonstrated by appropriate proof of identification.
2. Subjects will have a:

   2.1. BMI of 18.5 to 30.0 kg/m2, inclusive 2.2. body weight exceeding 52 kg (males) or 45 kg (females)
3. Subjects will be in good health, as judged by the PI or the appropriately qualified designee based on:

   3.1. medical history 3.2. physical examination 3.3. vital signs assessment 3.4. 12-lead ECG 3.5. clinical laboratory evaluations 3.6. lung function tests
4. Subjects will have given their written informed consent to participate in the study and will have agreed to abide by the study restrictions.
5. Subjects must demonstrate the ability to comprehend the informed consent form (ICF), be able to communicate well with the PI or the appropriately qualified designee, understand and comply with the requirements of the study, and be judged suitable for the study in the opinion of the PI or the appropriately qualified designee.
6. Subjects will be willing to refrain from consuming alcohol within 24 hours prior to Admission.
7. Subjects will be regular smokers of factory made, non-menthol cigarettes whose chosen brand is within the ISO tar bands 6 to 10 mg, inclusive and should not change their usual brand cigarette for the duration of the study.
8. Subjects will have smoked their chosen brand for a minimum of 6 months and will have smoked for at least 3 years prior to Screening, and will typically smoke at least 10 and a maximum of 30 CPD.
9. Subjects must have a urine cotinine level >200 ng/mL and an ECO measurement of >10 ppm at Screening.
10. Subjects will be willing to use the study products and smoke only the study products provided to them during clinical confinement and to abstain from smoking when required.

Exclusion Criteria:

1. Male subjects who do not agree, or whose partners of childbearing potential do not agree, to use a barrier method of contraception (i.e., a condom with spermicide) in addition to a second highly effective method of contraception used by their female partners or to refrain from donating sperm from Admission for Visit 1 until 5-7 days after Discharge.
2. Female subjects of childbearing potential who do not agree to use a highly effective method of birth control in conjunction with male barrier method contraception (i.e., a condom with spermicide) from the time of signing the ICF until 5-7 days after Discharge.
3. Female subjects who are pregnant or breastfeeding. This will be confirmed at Screening and at each Admission. Any female subject who becomes pregnant during this study will be withdrawn.
4. Subjects who have donated:

   4.1. ≥450 mL of blood within 90 days prior to Admission 4.2. plasma in the 7 days prior to Admission 4.3. platelets in the 6 weeks prior to Admission
5. Subjects who have an acute illness (e.g., upper respiratory tract infection, viral infection, etc.) requiring treatment within 4 weeks prior to Admission.
6. Subjects who have used any nicotine or tobacco product other than commercially manufactured non-menthol, filter cigarettes within 14 days of Screening.
7. Subjects who are self-reported non-inhalers (smokers who draw smoke from the cigarette into the mouth and throat but who do not inhale). Subjects who are determined as non-inhalers at Screening will be excluded.
8. Subjects who, prior to enrolment, are planning to quit smoking in the next 12 months of Screening. All subjects will be informed that they are free to quit smoking and withdraw from the study at any time. Any subject who decides to quit smoking will be directed to appropriate stop smoking services
9. Subjects who have a significant history of alcoholism or drug/chemical abuse within 24 months prior to Screening, as determined by the PI or the appropriately qualified designee.
10. Subjects who have a positive urine drugs of abuse or alcohol screen (confirmed by repeat) at Screening or Admission.
11. Subjects who:

    11.1. have serum hepatitis 11.2. are carriers of the hepatitis B surface antigen (HBsAg) 11.3. are carriers of the hepatitis C antibody 11.4. have a positive result for the test for human immunodeficiency virus (HIV) antibodies.
12. Subjects who have used prescription or OTC bronchodilator medication (e.g., inhaled or oral β-adrenergic agonists) to treat a chronic condition within the 12 months prior to the first Admission (Visit 1) and throughout the study.
13. Subjects who have received any medications or substances (other than tobacco) which:

    13.1. are known to be strong inducers or inhibitors of CYP enzymes within 14 days or 5 half-lives of the drug (whichever is longer) prior to the first Admission (Visit 1) and throughout the study.
14. Subjects who are planning to undergo significant lifestyle changes during the study e.g., big change in exercise levels.
15. Subjects who are unable to communicate effectively with the PI/study staff (i.e., language problem, poor mental development, or impaired cerebral function).
16. Subjects who are unwilling or unable to comply with the study requirements.
17. Employees, and immediate relatives, of the tobacco industry or the clinical site.
18. Subjects who are still participating in another clinical study (e.g., attending follow-up visits) or who have participated in a clinical study involving administration of an investigational drug (new chemical entity) in the past 3 months prior to first Admission (Visit 1).
19. Subjects who have any clinically relevant abnormal findings on the physical examination, medical history, ECG, lung function tests (forced expiratory volume in 1 second/ forced vital capacity [FEV1/FVC]), or clinical laboratory panel, unless deemed not clinically significant by the PI or the appropriately qualified designee.
20. Subjects who have, or who have had a history of, any clinically significant neurological, gastrointestinal, renal (including urinary tract infection or nephrolithiasis), hepatic, cardiovascular, psychiatric, respiratory, metabolic, endocrine, haematological or other major disorder that, in the opinion of the PI or the appropriately qualified designee, would jeopardise the safety of the subject or impact on the validity of the study results.
21. Subjects who have previously been diagnosed with any form of malignancy.
22. Subjects who have any clinically significant abnormal laboratory safety findings at Screening and prior to first product use, as determined by the PI or the appropriately qualified designee (1 repeat assessment is acceptable).
23. Subjects who have previously been randomised into or withdrawn from this study.
24. Subjects who, in the opinion of the PI or the appropriately qualified designee, should not participate in this study.

Compliance with all inclusion and exclusion criteria will be reaffirmed at each study Visit.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2017-12-08 (Actual)

PRIMARY OUTCOMES:
Cmax | -5, 1, 2, 3, 4, 5, 6, 7, 8, 15, 60, 120, 180 and 240 minutes in relation to the first puff
  To assess the maximum nicotine concentration when subjects smoke a single cigarette

SECONDARY OUTCOMES:
AUC0-last | -5, 1, 2, 3, 4, 5, 6, 7, 8, 15, 60, 120, 180 and 240 minutes in relation to the first puff
  To assess the area under the concentration curve from time 0 to last the time-point when subjects smoke a single cigarette
Tmax | -5, 1, 2, 3, 4, 5, 6, 7, 8, 15, 60, 120, 180 and 240 minutes in relation to the first puff
  To assess the time to maximum nicotine concentration when subjects smoke a single cigarette
Puff Volume | During the time required to smoke a single cigarette (up to 8 minutes)
  To assess puff volume when subjects smoke a single cigarette
Puff duration | During the time required to smoke a single cigarette (up to 8 minutes)
  To assess puff duration when subjects smoke a single cigarette
Number of puffs | During the time required to smoke a single cigarette (up to 8 minutes)
  To assess number of puffs when subjects smoke a single cigarette
Inhalation volume | During the time required to smoke a single cigarette (up to 8 minutes)
  To assess inhalation volume when subjects smoke a single cigarette
Exhalation volume | During the time required to smoke a single cigarette (up to 8 minutes)
  To assess exhalation volume when subjects smoke a single cigarette

CONTACTS AND LOCATIONS:
Overall Officials: Johnston Stewart, MB, Principal Investigator — Celerion GB Ltd
Locations (1):
- Celerion, Belfast, Northern Ireland, United Kingdom